CLINICAL TRIAL: NCT00045448
Title: Single Center Open-Label Non-Comparative Phase I Dose Finding Study Of Weekly Flavopiridol In Combination With Weekly Docetaxel In Patients With Advanced Solid Tumors
Brief Title: Combination Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: AVENTIS-HMR1275A/1501; MSKCC-02034; NCI-G02-2106; CDR0000256563 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2009-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — alvocidib; Docetaxel

INTERVENTIONS:
Drug: alvocidib
Drug: docetaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining flavopiridol with docetaxel in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of flavopiridol when administered in combination with 2 different doses of docetaxel in patients with advanced solid tumors.
* Determine the clinical pharmacokinetics of this regimen in these patients.
* Determine, preliminarily, the therapeutic activity of this regimen in these patients.

OUTLINE: This is a dose-escalation study of flavopiridol.

Patients receive docetaxel IV over 30 minutes followed at least 4 hours later by flavopiridol IV over 1 hour on days 1, 8, and 15. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of flavopiridol until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Separate MTDs of flavopiridol are determined when flavopiridol is combined with 2 different doses of docetaxel. A total of 10 patients are treated at each flavopiridol MTD.

Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-56 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced solid tumor that is refractory to standard therapy or for which no standard therapy exists
* Measurable or evaluable disease
* No symptomatic or untreated CNS metastases or primary CNS neoplasm

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 70-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3
* Hemoglobin at least 8 g/dL

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)
* SGOT/SGPT no greater than 2.5 times ULN if alkaline phosphatase no greater than ULN OR
* Alkaline phosphatase no greater than 2.5 times ULN if SGOT/SGPT no greater than ULN

Renal

* Creatinine no greater than 1.5 mg/dL

Cardiovascular

* No history of cardiac arrhythmias
* No congestive heart failure
* No myocardial infarction within the past 6 months

Other

* No concurrent serious or uncontrolled infection
* No diabetes not adequately controlled with medication
* No peripheral neuropathy greater than grade 1
* No known allergy to docetaxel or other medications formulated in Polysorbate 80
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 4 weeks since prior immunotherapy

Chemotherapy

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Prior taxanes allowed
* No prior flavopiridol

Endocrine therapy

* At least 4 weeks since prior hormonal therapy

Radiotherapy

* At least 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* Recovered from prior therapy
* No prior enrollment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2006-01 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary K. Schwartz, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States